CLINICAL TRIAL: NCT02675699
Title: Effectiveness of an Implementation Optimisation Intervention Aimed at Increasing Parent Engagement in HENRY, a Childhood Obesity Prevention Programme: a Cluster Randomised Controlled Trial
Brief Title: The Optimising Family Engagement in HENRY (OFTEN) Study
Acronym: OFTEN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Leeds (Other)
Responsible Party: Principal Investigator, Maria Bryant, NIHR Career Development Fellow, University of Leeds
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: RG.AUHE.102510
Record Dates: First submitted 2016-01-28; First posted 2016-02-05 (Estimated); Last update posted 2022-03-25 (Actual); Status verified 2019-07

CONDITIONS: Childhood Obesity
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Optimisation + HENRY (Experimental)
  Interventions: Behavioral: Optimisation + HENRY
- HENRY as standard (Active Comparator)
  Interventions: Behavioral: HENRY as standard

INTERVENTIONS:
Behavioral: Optimisation + HENRY — HENRY HENRY is an 8-week childhood obesity prevention programme delivered in Children's Centres in the UK by trained practitioners, aiming to provide parents with skills and knowledge to support healthy lifestyles in preschool children and their families. The programme aims to build parents' skills, knowledge and confidence to change old habits and provide healthier nutrition.
  OPTIMISATION A tailored 'Optimisation' intervention has being developed to support local authorities and Children's Centres to promote HENRY implementation, based on an ethnography of Children Centres, including interviews with staff and other stakeholders and input from parents. Development was underpinned by strong theories of behaviour change and will be guided by the intervention planning framework; the Behaviour Change wheel using a systematic approach. Strategies have been developed to improve parent motivation to enrol on to HENRY and promote parent self-efficacy to continue to attend.
  Arms: Optimisation + HENRY
Behavioral: HENRY as standard — Local Authorities / Children's Centres that are assigned to the control group will continue with standard HENRY practice. Current HENRY QA practice involves the review of process data by HENRY central office with provision of written and oral feedback. This will continue in both trial arms and will be monitored.
  Arms: HENRY as standard

SUMMARY:
This study will test whether parent engagement (recruitment, attendance) in a Childhood obesity prevention programme (HENRY) can be improved in local authorities randomised to receive an Optimisation intervention (in addition to standard HENRY) compared to those continuing to deliver the programme as standard.

DETAILED DESCRIPTION:
BACKGROUND: Rising rates of obesity in preschool children are alarming and emphasise the need for evidence-based approaches to prevent obesity, which can be successfully implemented in communities. Although robust, theory-based prevention programmes exist, it is often a challenge to get parents to attend them and adopt positive behaviour changes in their families.

AIM: To evaluate the effectiveness of a recently developed 'Optimisation intervention' to optimise parent engagement in a community based obesity prevention programme 'HENRY', using routinely collected process data from existing sites commissioned to deliver HENRY in the UK

DESIGN: Multi-centre, cluster randomised controlled trial. As research will judge the ability of local authorities and their Centres to optimise implementation of HENRY, a cluster randomised design, has been chosen with local authority as the unit of randomisation. Local authorities will be randomised in a 1:1 allocation ratio (HENRY+ Optimisation Intervention; HENRY alone control) by a statistician at Leeds CTRU, using minimisation algorithm with random element, stratifying on baseline level of implementation (proportion of Centres meeting none of the 2 primary outcome implementation criteria/ meeting 1 or 2 of the criteria)) size of local authorities (number of Children's Centres (< 10/ ≥10)) and area deprivation (≤10% />10% ranking within Index of Multiple Deprivation at the Lower Layer Super Output Area).

Consent to participate will be sought at the cluster level (local authorities) and from the Centres within each local authority using an opt-out approach.

CONTROL ARM: HENRY delivered as standard. HENRY (Health, Exercise, Nutrition for the Really Young) is an 8-week programme delivered in Children's Centres (CCs), aiming to provide parents with skills and knowledge to support healthy lifestyles in preschool children and their families. It was set up in 2006 with Department of Health support aimed at reversing rising trends in school entry age obesity. HENRY is currently delivered in 32 local areas across England and Wales by trained health and community practitioners.

ACTIVE ARM: HENRY as standard plus an optimisation intervention to enhance parent engagement (recruitment and attendance) in the 8 week programme. A tailored 'Optimisation' intervention has been developed with a NIHR funds (CDF 2014-07-052) to support local authorities and Children's Centres to promote HENRY implementation, based on observations of positive deviants, interviews with Children Centre staff and other stakeholders, and input from parents. The resulting optimisation package is a multi-component intervention implemented at multi-levels (local authorities, Centres, parents). Precise details can not currently be disclosed to do risk of contamination.

ANALYSIS: Primary outcome analysis will be on the intention-to treat Population using a 3-level hierarchical model, with courses (or participants) nested within CCs within LA, adjusting for randomization minimisation variables. Differences in parent engagement, corresponding 95% CI, p-values and ICCs will be reported.

ELIGIBILITY:
Inclusion Criteria:

Local authorities:

* Local authorities providing data from at least 4 Children's Centres
* Courses delivered by trained staff who have been certified by HENRY

Children's Centres:

* At least one course to be delivered per Centre per year
* Sites with a history of providing process data for the previous year.

There will be no exclusions based on the demographics of Children's Centres, but location will be monitored to ensure inclusion of those with diverse social and environmental characteristics.

-

Exclusion Criteria:

Local authorities:

* Areas which have plans to decommission the HENRY intervention during the course of the trial; or who are not planning on running HENRY programmes during the trial period.

Children's Centres:

* Centres where ethnography has taken place during Study 2
* Centres who are not planning on running HENRY programmes during the trial period

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Number of parents engaging with the HENRY programme measured using Centre level process data | 12 month post randomisation (allowing 3 months for Optimisation intervention implementation and collecting data from 1- 2 HENRY courses per site).
  Centre level data: A combined outcome of parent engagement based on the number of parents recruited per course and the attendance rate. In order to be effective, courses need improve parent engagement and retain parents to continue on the course.

SECONDARY OUTCOMES:
Level of parent compliance to HENRY content measured via self-reported changes in frequency that fruits and vegetables are consumed each day by infants | 12 months post randomisation
  Compliance will be measured using a proxy of parent reported frequency of consumption of fruits /vegetables by children/ day/ course. This will be assessed at the parent-level as a binary variable
Parenting self-efficacy | 12 months post randomisation
  Adapted Parenting Self-Agency Measure
  Parenting self-agency measure (Dumka 1996)
Eating behaviours | 12 months post randomisation
  Golan (1998) Family Eating and Activity Habits Questionnaire
Family activity | 12 months post randomisation
  Bespoke HENRY brief activity questionnaire
Daily intake of key indicator foods in infants | 12 months post randomisation
  Modified validated Food Frequency Questionnaire (Hammond 1993)

OTHER OUTCOMES:
Cost effectiveness measured using acceptability curves | 12 months post randomisation
  Economic evaluation of the Optimisation intervention. Commissioner willingness to pay for the Optimisation Intervention. The true value of the optimised intervention will be ascertained following discussions with the commissioners to determine their willingness to pay. Recruitment and attrition will be categorised as achieved or not (binary) at the centre-level, although continuous data will also be provided to aid commissioners discussion from the willingness to pay analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Medicine and Health, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Data IP is held with the HENRY organisation

REFERENCES:
- [Result] Bryant M, Burton W, Collinson M, Farrin A, Nixon J, Stevens J, Roberts K, Foy R, Rutter H, Copsey B, Hartley S, Tubeuf S, Brown J. A cluster RCT and process evaluation of an implementation optimisation intervention to promote parental engagement enrolment and attendance in a childhood obesity prevention programme: results of the Optimising Family Engagement in HENRY (OFTEN) trial. Trials. 2021 Nov 5;22(1):773. doi: 10.1186/s13063-021-05757-w. PMID 34740373
- [Derived] Bryant M, Burton W, Cundill B, Farrin AJ, Nixon J, Stevens J, Roberts K, Foy R, Rutter H, Hartley S, Tubeuf S, Collinson M, Brown J. Effectiveness of an implementation optimisation intervention aimed at increasing parent engagement in HENRY, a childhood obesity prevention programme - the Optimising Family Engagement in HENRY (OFTEN) trial: study protocol for a randomised controlled trial. Trials. 2017 Jan 24;18(1):40. doi: 10.1186/s13063-016-1732-3. PMID 28115006

DOCUMENTS (1):
  • Study Protocol (2016-02-04): https://cdn.clinicaltrials.gov/large-docs/99/NCT02675699/Prot_000.pdf